CLINICAL TRIAL: NCT04226105
Title: An Open-label, Randomized, Multi-center, Parallel-group Clinical Trial Comparing the Efficacy and Safety of GP40081 (OOO "GEROPHARM", Russia) Compared to NovoMix® 30 FlexPen® (Novo Nordisk A/S, Denmark) in Type 2 Diabetes Mellitus Patients
Brief Title: Efficacy and Safety of GP40081 Сompared to NovoMix® 30 FlexPen® in Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP40081-P4-31
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP40081 (Experimental): Subcutaneous (SC), up to Week 26
  Interventions: Drug: GP40081
- NovoMix® 30 FlexPen® (Active Comparator): Subcutaneous (SC), up to Week 26
  Interventions: Drug: NovoMix 30

INTERVENTIONS:
Drug: GP40081 — 1 ml of the GP40081 contains 100 units soluble insulin aspart/protamine-crystallised insulin aspart in the ratio 30/70. Insulin aspart 30 mix is self-administered drug by SC injection 1-3 times per day before meal intake.
  Other Names: Insulin aspart 30 mix
  Arms: GP40081
Drug: NovoMix 30 — 1 ml of the NovoMix 30 contains 100 units soluble insulin aspart/protamine-crystallised insulin aspart in the ratio 30/70. Insulin aspart 30 mix is self-administered drug by SC injection 1-3 times per day before meal intake.
  Other Names: Insulin aspart 30 mix
  Arms: NovoMix® 30 FlexPen®

SUMMARY:
This trial is a multi-center, open-label, randomized, parallel group trial in adult patients with T2DM comparing the efficacy and safety of GP40081 (insulin asapart mix 30, GEROPHARM) with that of NovoMix® 30 FlexPen®.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Diabetes mellitus type 2 for at least 6 months before the screening (WHO criteria 1999-2013).
* Glycated haemoglobin (HbA1c) level of 7.6 to 12.0 % at screening (both values inclusive).
* Indications for exogenous insulin therapy.
* Body mass index (BMI) of 18.5 to 40 kg/m2 at screening (both values inclusive).
* Insulin-naive patients or prior insulin therapy at least 6 months before randomization.
* The subject is able and willing to comply with the requirements of the study protocol

Exclusion Criteria:

* Contraindication to the use of insulin aspart 30 mix.
* History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the trial, OR history of significant allergic drug reactions.
* History of severe hypoglycemia for 6 months before the screening.
* History of severe hyperglycemia for 6 months before the screening.
* Bariatric surgery for 12 months to screening.
* Glucagon-like peptide-1 (GLP-1)-based therapies for 8 weeks to screening.
* Insulin resistance over 1.5 U/kg insulin pro day.
* Change INN of insulin for 6 months before the randomisation.
* History of treatment any experimental drugs or medical devices for 3 months before the randomisation.
* Presence of severe diabetes complications.
* Night work.
* History of administration of glucocorticoids (14 days or more) for 1 year before the screening.
* Administration of any immunosuppressive drugs (Cyclosporinum, Methotrexate, Rituximab, etc.).
* History of vaccination for 6 months before the randomisation.
* History of autoimmune disease, except vitiligo and controlled autoimmune polyglandular syndrome (APS) types 1-3, except vetiligo and Hashimoto's thyroiditis.
* Pregnant and breast-feeding women.
* Deviation of the laboratory results conducted during the screening: Hemoglobin value < 9,0 g/dl; Hematocrit value < 30 %; ALT and AST value > 2 folds or ALT or AST value > 3 folds as high as maximal normal value; Serum bilirubin value > 2 folds as high as maximal normal value (except Gilbert's syndrome).
* History of haematological disorders that can affect the reliability of HbA1c estimation (haemoglobinopathies, hemolytic anaemia, etc.).
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B (HbSAg), hepatitis C (HCVAb) or syphilis (Treponema pallidum) antibodies at the screening.
* Acute inflammation disease for 3 weeks before the screening.
* History of unstable angina, myocardial infarction, severe arrhythmia, heart failure III or IV NYHA for 1 year before the screening.
* History of stroke or TIA for 6 months before the screening.
* Serious blood loss for 3 months before the screening (blood donation, surgery procedure, etc.).
* The inability of the patient to assess their condition because of mental or physical disorders.
* History of drug, alcohol abuse for 3 years before the screening.
* History of oncology disorders for 5 years before the screening.
* History of transplantation, except 3 months after a corneal transplant.
* History or presence of a medical condition or disease that in the investigator's opinion would embarrass glycemic control and completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | 26 weeks
  Change from baseline in titer of antibodies to human insulin

SECONDARY OUTCOMES:
Glycated hemoglobin | 26 weeks
  Change in HbA1c from baseline
Adverse Events frequency and degree | 26 weeks
  Hypoglycemic episodes (glucose level < 3.9 mmol/l) frequency; Occurrence of local reactions at injection sites; Occurrence allergic reactions
Fasting Plasma Glucose Level | 26 weeks
  Change in fasting plasma glucose level from baseline
Seven-Point Glucose Testing | 22 weeks
  Change in seven-point glucose testing results from baseline
Total Insulin Dose | 22 weeks
  Change in total insulin dose per body weight (U/kg) from baseline
Body Mass Index | 26 weeks
  Change in BMI from baseline
Treatment Satisfaction: The Diabetes Treatment Satisfaction Questionnaire | 26 weeks
  Change in treatment satisfaction from baseline. Questions 1, 4, 5, 6, 7 and 8 assesses treatment satisfaction (summed these 6 questions). Questions 2 and 3 assess the burden from hyper- and hypoglycemia. DTSQ is The Diabetes Treatment Satisfaction Questionnaire, scored from 0-36 points with higher scores indicating better satisfaction.
Achievement of Glycated Hemoglobin Goals | 26 weeks
  The frequency of achievement glycated hemoglobin goals
Achievement of Glycated Hemoglobin < 7% | 26 weeks
  The frequency of achievement glycated hemoglobin < 7% ( 7% inclusive)

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Kazan Endocrinology Dispensary, Kazan'
  - Krasnoyarsk State Medical University named after Professor V.F. Voino-Yasenetsky, Krasnoyarsk
  - V.A. Baranov Republic Hospital, Petrozavodsk
  - City Diagnostic Center № 1, Saint Petersburg
  - City Hospital № 2, Saint Petersburg
  - City Polyclinic № 117, Saint Petersburg
  - EosMed, Saint Petersburg
  - Institute of Medical Research, Saint Petersburg
  - Research Center Eco-Safety, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Diabetes Center, Samara
  - Volgograd Region Clinical Hospital №1, Volgograd

IPD SHARING:
Plan to Share IPD: No